CLINICAL TRIAL: NCT00716742
Title: Safety and Efficacy Study of Bimatoprost, Latanoprost, and Travoprost in Patients With Elevated Intraocular Pressure (IOP) and Open-angle Glaucoma (OAG)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro2
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Results first posted 2012-01-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2011-11

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Latanoprost; Travoprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: bimatoprost 0.03% latanoprost 0.005% travoprost 0.004%
  Interventions: Drug: bimatoprost 0.03%, latanoprost 0.005%, and travoprost 0.004%

INTERVENTIONS:
Drug: bimatoprost 0.03%, latanoprost 0.005%, and travoprost 0.004% — 1 drop in eye(s) every evening
  Other Names: Lumigan®; Xalatan®; Travatan®

SUMMARY:
To investigate the effectiveness of the newer IOP-lowering therapies, as prescribed in normal clinical practice, in larger patient numbers. Patients will be assessed at baseline, at each follow-up visit (follow-up visits are variable as per physician discretion) and at final follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Primary Open-Angle Glaucoma or Ocular Hypertension newly diagnosed OR presenting with insufficiently controlled IOP on current medication (in the opinion of the treating physician)
* Patient is having both eyes treated

Exclusion Criteria:

* Contraindications per product labelling will apply.
* Patients with any ophthalmic co-morbidity with an influence on visual field deterioration or optic nerve head damage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients can be either: (a) newly diagnosed and require, in the judgment of the treating physician, one of study agents as first-line treatment, (b) have an insufficiently controlled IOP on their current medication (any but not more than two in combination), and a treatment switch to one of study agents is an acceptable option.
Sampling Method: Non-Probability Sample
Enrollment: 1099 (Actual)
Dates: Start 2004-09; Primary Completion 2007-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Murfreesboro, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lumigan®: bimatoprost 0.03%
- Travatan®: travoprost 0.004%
- Xalatan®: latanoprost 0.005%
Period: Baseline
Arm/Group | Lumigan® | Travatan® | Xalatan®
Started | 364 | 370 | 365
Completed | 347 | 356 | 352
Not Completed | 17 | 14 | 13
Period: 1 Year Follow-up
Arm/Group | Lumigan® | Travatan® | Xalatan®
Started | 347 | 356 | 352
Completed | 160 | 163 | 152
Not Completed | 187 | 193 | 200
Period: 2 Year Follow-up
Arm/Group | Lumigan® | Travatan® | Xalatan®
Started | 160 | 163 | 152
Completed | 56 | 67 | 50
Not Completed | 104 | 96 | 102
Period: 3 Year Follow-up
Arm/Group | Lumigan® | Travatan® | Xalatan®
Started | 56 | 67 | 50
Completed | 26 | 35 | 29
Not Completed | 30 | 32 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumigan® | Travatan® | Xalatan® | Total
Number analyzed (Participants) | 364 | 370 | 365 | 1099
Age Continuous [Median (Full Range); unit: years] | 65.5 [21 to 97] | 67.0 [32 to 98] | 67.0 [23 to 95] | 67.0 [21 to 98]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 206 | 201 | 617
  Male | 154 | 164 | 164 | 482

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bilateral Intraocular Pressure (IOP) at One Year
Description: Change from baseline in bilateral (both eyes) IOP at the 1 year follow-up visit. IOP is a measure of the fluid pressure inside the eye. The bilateral IOP was calculated as an average between both eye's IOP. A negative number change from baseline indicates reduction in IOP (improvement).
Time Frame: Baseline, 1 Year
Population: Intent-to-treat, which includes all patients who started the study and completed the one-year follow-up visit and whose data was available for this outcome measure.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Lumigan® | Travatan® | Xalatan®
Number analyzed (Participants) | 160 | 162 | 152
Millimeters of mercury (mmHg)
  Baseline | 20.8 (5.2) | 20.3 (5.0) | 20.6 (5.2)
  Change from Baseline at 1 Year | -4.8 (3.3) | -4.3 (2.7) | -4.3 (2.9)

ADVERSE EVENTS:
Arm/Group | Lumigan® | Travatan® | Xalatan®
Serious Adverse Events (participants affected / at risk) | 5/364 | 2/370 | 6/365
Other Adverse Events (participants affected / at risk) | 0/364 | 0/370 | 0/365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lumigan® (N=364) | Travatan® (N=370) | Xalatan® (N=365)
Death (General disorders) | 5 | 2 | 6 — Causes of Death not specified

LIMITATIONS AND CAVEATS:
Data for 2-year and 3-year follow-up not interpretable due to extremely high drop out rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.